CLINICAL TRIAL: NCT00050700
Title: Muscarinic Cholinergic Receptor Imaging in Depression
Brief Title: Brain Imaging in Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030001; 03-M-0001
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-14

CONDITIONS: Depression; Bipolar Disorder
Keywords: PET; [18F]FP-TZTP; Bipolar Disorder; Major Depressive Disorder; Muscarinic 2 Receptors
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder, Major

SUMMARY:
The purpose of this study is to use brain imaging technology to examine the role of certain brain receptors and the nervous system chemical acetylcholine in major depression.

The cholinergic system involves the regulation of neurotransmitters and the brain receptors to which they bind. Evidence suggests that the cholinergic system may play a role in the development of depression. Acetylcholine is a neurotransmitter that binds to certain brain receptors called muscarinic cholinergic receptors. Cholinomimetic drugs (drugs that stimulate the cholinergic system) often exacerbate depressive symptoms in people with mood disorders and in healthy individuals. This increase in depressive symptoms may be caused by stimulation of muscarinic acetylcholine receptors (mAChRs), but further study is needed to confirm this. This study will use positron emission tomography (PET) and magnetic resonance imaging (MRI) to study the function of mAChRs in individuals with depression.

Participants in this study will undergo a physical examination, psychiatric interviews, neuropsychological tests, PET and MRI scans, and rating scales of depression, anxiety, and negative thinking symptoms. Questions about behavior and functioning will be asked and blood samples will be collected for genetic analysis.

DETAILED DESCRIPTION:
Several paths of evidence converge in implicating a role for the cholinergic system in the pathophysiology of affective illness. In both unipolar depressed and euthymic bipolar subjects, cholinomimetic drugs (i.e., muscarinic agonists, acetylcholinesterase inhibitors) exacerbate depressive signs and symptoms such as dysphoria, psychomotor retardation, impairment of attention and memory, hypothalamic pituitary adrenal axis hyperactivity and sleep EEG abnormalities. In healthy subjects, the acetylcholinesterase inhibitor physostigmine elicits a range of depressive symptoms including dysphoria, anergia, psychomotor slowing, emotional lability, sleep disturbances, memory and concentration impairment, and with higher doses, tearfulness and depression. These effects have been shown to reflect stimulation of muscarinic receptors. Cholinomimetics also exacerbate behavioral despair in putative animal models of depression. Conversely, the anticholinergic agent biperidine improved symptoms of depression in a placebo controlled study. Moreover, muscarinic cholinomimetics and a choline rich nutrient, lecithin (phosphatidylcholine) exert antimanic effects in bipolar subjects.

Potentially consistent with these observations, depressed subjects exhibit hypersensitivity to cholinomimetic agents. Administration of muscarinic cholinergic agonists, ACh releasing agents or acetylcholinesterase inhibitors induce exaggerated effects on REM density and latency in depressed subjects than in healthy controls. In addition, both manic and depressed bipolar subjects show increased pupillary sensitivity to the muscarinic cholinergic agonist pilocarpine relative to controls.

Despite the data implicating the mAChR receptor system in mood disorders, no direct in vivo investigations of the central mAChR have been performed in depressed subjects. A novel PET radioligand, [(18)F]FP-TZTP was recently developed by Eckelman as a selective agonist of M(2) receptors. Because the M(2) receptor functions predominately as a presynaptic release-controlling autoreceptor, decreased distribution volume (V) of this receptor could conceivably give rise to increased postsynaptic muscarinic receptor sensitivity.

This application proposes a pilot PET study of M(2) receptor distribution volume in currently depressed subjects with major depressive disorder (n=30), currently depressed subjects with bipolar disorder (n=30), and psychiatrically healthy controls (n=30). The proposed pilot study will test the central hypothesis that M(2) receptor V is decreased in regions where they are primarily located presynaptically in depressed subjects relative to healthy controls. The proposed study will advance knowledge regarding the pathophysiology of depression.

ELIGIBILITY:
* INCLUSION CRITERIA - MDD Depressed Sample:

Thirty subjects (ages 18-45) male and female will be selected, with primary MDD currently depressed as defined by DSM-IV criteria for recurrent MDD and current HDRS score in the moderately-to-severely depressed range (greater than 18) and who have a first degree relative with MDD but no first degree relatives with mania, alcoholism, or antisocial personality disorder.

INCLUSION CRITERIA - Bipolar Depressed Sample:

Thirty subjects (ages 18-45) male and female will be selected who meet DSM-IV criteria for bipolar I or II disorder and are currently depressed, with HDRS score in the moderately-to-severely depressed range (greater than 18). Subjects may be inpatients or outpatients. Because effective treatment will not be discontinued for the purposes of this protocol, subjects will be identified who have never been treated or who have discontinued medication due to lack of efficacy, noncompliance, physician order, or other reasons prior to study entry.

INCLUSION CRITERIA - Healthy, Control Sample:

Thirty subjects (ages 18-45) male and female who have not met criteria for any major psychiatric disorder will be selected. From this large sample a control subject will be matched to each depressed subject for age, gender, handedness and stage of menstrual cycle. The control subjects will have no known first degree relatives with mood disorders.

EXCLUSION CRITERIA:

Subjects must not have taken antidepressant or other medications likely to alter monoamine neurochemistry or cerebrovascular function for at least 3 weeks (8 weeks for fluoxetine and for any drug with known anticholinergic effects) prior to scanning. Because effective medications will not be discontinued for the purposes of this study, subjects will be identified who have never been treated or who have discontinued medication due to lack of efficacy, noncompliance, physician order or other reasons prior to study entry. Subjects will also be excluded if they: a) serious suidical ideation or behavior - 1) thoughts of suicide within the past three months which are accompanied by intet to harm oneself, serious consideration of means or plan to attempt suicide, evidence of arranging for a suicide attemp (e.g. giving away prized possessions, updating a will) or clear desire to commit suicide; 2) suicide attempts within the previous one year; or 3) a current plan to inflict self harm or physical evidence suspicious for having engaged in a suicide attempt.

Subjects will also be excluded if they had any significant comorbid condition in the last year, c) psychosis to the extent that the ability to provide informed consent is in doubt, d) history of any major psychiatric disorder (other than the target mood disorder) arising temporally before the initial mood episode, e) medical or neurological illnesses (i.e. seizure disorder, a coma in past) likely to affect physiology or anatomy, f) a history of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria), g) are HIV positive or have AIDS, h) current pregnancy (documented by history and pregnancy testing prior to scanning), i) current breast feeding, j) general MRI exclusion criteria which include the subject having a pacemaker or significant claustrophobia and k) if they are smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2002-12-16; Study Completion 2010-05-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Allen TG. The role of N-, Q- and R-type Ca2+ channels in feedback inhibition of ACh release from rat basal forebrain neurones. J Physiol. 1999 Feb 15;515 ( Pt 1)(Pt 1):93-107. doi: 10.1111/j.1469-7793.1999.093ad.x. PMID 9925881
- [Background] Arango V, Underwood MD, Boldrini M, Tamir H, Kassir SA, Hsiung S, Chen JJ, Mann JJ. Serotonin 1A receptors, serotonin transporter binding and serotonin transporter mRNA expression in the brainstem of depressed suicide victims. Neuropsychopharmacology. 2001 Dec;25(6):892-903. doi: 10.1016/S0893-133X(01)00310-4. PMID 11750182
- [Background] Baratti CM, Opezzo JW, Kopf SR. Facilitation of memory storage by the acetylcholine M2 muscarinic receptor antagonist AF-DX 116. Behav Neural Biol. 1993 Jul;60(1):69-74. doi: 10.1016/0163-1047(93)90742-z. PMID 8216161